CLINICAL TRIAL: NCT02764203
Title: ChOcolate COnsumption And Blood Pressure (COCOA-BP): A Wearable Devices Pilot Trial
Acronym: COCOA-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S2363
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Health Behavior; Blood Pressure
Keywords: Dark Chocolate; Blood Pressure; Wearable Devices; Digital Health
MeSH Terms: conditions — Health Behavior | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chocolate consumption (Experimental): Subjects will consume 50g of dark chocolate for 2 weeks and have their blood pressure compared before chocolate and after chocolate
  Interventions: Other: Dark Chocolate; Device: Wearable devices

INTERVENTIONS:
Other: Dark Chocolate — 50g dark chocolate consumed for a period of 2 weeks
Device: Wearable devices — Up to three wearable devices will be worn by the subject to measure parameters such as heart rate, blood pressure and number of steps

SUMMARY:
The COCOA-BP Trial is designed to assess the impact of 50g daily dark chocolate intake on blood pressure and compare outcome data derived from wearable/digital health devices to data derived from standard methods. Additionally, the usability of the wearable technology will be evaluated.

DETAILED DESCRIPTION:
The COCOA-BP Trial is a prospective, single-center, single-arm, Boston Scientific volunteer trial, designed to assess the impact of 50g daily dark chocolate intake on blood pressure and compare outcome data derived from wearable/digital health devices to data derived from standard methods. Additionally, the usability of the wearable technology will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject has an iPhone (5 or higher)
* Subject is willing to comply with all trial requirements
* Subject understands the trial requirements and procedures and provides written informed consent before any trial-specific procedures are performed

Exclusion Criteria:

* Anyone part of the study execution team cannot be part of the trial
* Current smoker or history of smoking in the last 5 years (including E-cigarettes)
* Diabetes mellitus including those managed by diet alone
* Medically treated hypertension
* Diagnosed with persistent or frequent irregular heart beat (e.g. atrial flutter, atrial fibrillation)
* Permanent pacemaker or defibrillator implanted
* Subject is a women who is pregnant
* Known allergy to chocolate or cacao products
* Known allergy to skin adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Change in resting systolic blood pressure after daily dark chocolate | 14 days after daily consumption of dark chocolate

SECONDARY OUTCOMES:
Correlation of physical activity (steps) to resting blood pressure and heart rate | daily, for four weeks
Comparison of blood pressure derived from wearable digital health devices to data derived from standard methods | End of week two and end of week four
Comparison of heart rate derived from wearable digital health devices to data derived from standard methods | End of week two and end of week four

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Christen, MD, PhD, Principal Investigator — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: Undecided